CLINICAL TRIAL: NCT03810066
Title: Exploring the Theragnostic Value of Osimertinib in EGFR-mutated Lung Cancer (THEROS) - A Multicentric Phase II Study in Patients With TKI-resistant EGFR-mutated Lung Cancer Exhibiting Early Metabolic Response to Osimertinib
Brief Title: Exploring the Theragnostic Value of Osimertinib in EGFR-mutated Lung Cancer (THEROS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THEROS
Record Dates: First submitted 2019-01-10; First posted 2019-01-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: NSCLC; EGFR T790M; FDG-PET
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Simon 2 step design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — All patients will be treated with osimertinib 80 mg/d for one cycle (28 days).

SUMMARY:
This is a single arm, open label, multicentric proof-of-concept, phase II study in patients with EGFR-mutated non-small-cell lung cancer (NSCLC) with acquired TKI resistance who are "unknown" for EGFR T790M status due to non-informative or unfeasible tumor rebiopsy, and a negative finding for EGFR T790M in a standard plasma genotyping assay. All patients will receive osimertinib as continuous oral treatment for one cycle (28 days). Patients who demonstrate a metabolic response by FDG-PET scanning (to be conducted between day 15 and day 28 of cycle 1) will continue treatment until clinical or radiological progression. Osimertinib treatment will be terminated in patients not experiencing a metabolic response.

Primary objective:

To study the rate of early metabolic responses to osimertinib in patients with EGFR-mutated NSCLC and acquired TKI resistance who are "unknown" for EGFR T790M status due to non-informative or unfeasible tumor rebiopsy, and a negative finding for EGFR T790M in a standard plasma genotyping assay.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients (male/female) must be > 18 years of age.
3. EGFR-mutated NSCLC not amenable to curative treatment (surgery, curative radiochemotherapy).
4. Acquired resistance to a first- or second-generation EGFR-TKI (e.g. afatinib, erlotinib, gefitinib) following initial benefit (defined as objective response, or stable disease for at least 3 months)
5. No tumor rebiopsy available or negative result for EGFR T790M mutation status by a SoC molecular pathology test (e.g. Sanger sequencing, PCRbased genotyping, deep sequencing) of a rebiopsy of a progressive tumor lesion
6. Negative finding from EGFR T790M mutation testing in plasma-derived DNA using a SoC assay (e.g. Roche Cobas)
7. At least one tumor lesion with significant FDG uptake as determined by PET/CT scanning prior to study treatment
8. Consent to the research use of donated biological samples.
9. World Health Organization (WHO) performance status 0-2.
10. Patients must have a life expectancy ≥ 12 weeks.
11. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of childbearing potential, which will be repeated on a monthly basis, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
12. Male patients should be willing to use barrier contraception (see Restrictions, Section 3.6).
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. EGFR-mutated NSCLC and demonstration of the T790M resistance mutation by standard assay technology in tumor-derived or plasma-derived DNA
2. Absence of a tumor lesion with significant FDG uptake at PET/CT scanning prior to study treatment
3. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site)
4. Previous treatment with osimertinib or any experimental or approved mutationspecific EGFR-TKI with clinical activity against the EGFR T790M resistance mutation
5. Treatment with an investigational drug within one week or five drug half-lives (whichever is longer) of the compound (3 weeks for antibodies)
6. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 week prior) (Appendix A - Guidance regarding Potential Interactions With Concomitant Medications). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4. A list for drug interaction potential is found in section 5.1.6.4 of the osimertinib IB.
7. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study Treatment with the exception of alopecia and grade 2, prior chemotherapy related neuropathy.
8. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
9. Patients with symptomatic CNS metastases who are neurologically unstable
10. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
11. Fasting blood glucose levels above 150 mg/dl (precluding informative FDGPET/ CT scanning)
12. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    Absolute neutrophil count <1.5 x 109/L Platelet count <100 x 109/L Haemoglobin <90 g/L Alanine aminotransferase >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
13. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec obtained from the screening clinic ECG machine-derived QTc value
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including serum/plasma potassium level below lower level of normal), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
14. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
15. History of hypersensitivity to osimertinib (or drugs with a similar chemical structure or class to osimertinib) or any excipients of these agents
16. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
17. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of metabolic responses | 28 days
  Rate of metabolic responses as detected by FDG-PET before end of cycle 1. One cycle is defined as 28 days continuous treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. med. Martin Schuler, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Schuler M, Hense J, Darwiche K, Michels S, Hautzel H, Kobe C, Lueong S, Metzenmacher M, Herold T, Zaun G, Laue K, Drzezga A, Theegarten D, Nensa F, Wolf J, Herrmann K, Wiesweg M. Early Metabolic Response by PET Predicts Sensitivity to Next-Line Targeted Therapy in EGFR-Mutated Lung Cancer with Unknown Mechanism of Acquired Resistance. J Nucl Med. 2024 Jun 3;65(6):851-855. doi: 10.2967/jnumed.123.266979. PMID 38575188
- See also: Early Metabolic Response by PET Predicts Sensitivity to Next-Line Targeted Therapy in EGFR-Mutated Lung Cancer with Unknown Mechanism of Acquired Resistance — https://pubmed.ncbi.nlm.nih.gov/38575188/